CLINICAL TRIAL: NCT03517774
Title: Improving Prosthetic Care for Patients With a Lower Limb Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MaRS 3D-Printing
Record Dates: First submitted 2018-02-15; First posted 2018-05-07 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D Printed Socket (Experimental): All participants will received a 3D Printed Prosthetic
  Interventions: Device: 3D Printed Socket

INTERVENTIONS:
Device: 3D Printed Socket — Twenty participants will be fitted with a 3D Printed socket created using 3DPrintAbility hardware and software. To do this, a 3D model of the participants residual limb will be generated which will be used to create the 3D printed sockets. These 20 participants will also receive standard care for prosthetic fitting at SJR. The fittings will be done by one prosthetist. Our team will compare the feasibility, function, quality and stability of the prosthetics through quantitative, economic and qualitative analyses. All fittings will be done under the supervision of a qualified Sunnybrook prosthetist who has previous experience with using 3D printed technologies for creation of prosthetics.

SUMMARY:
Adults with lower limb amputation undergo rehabilitation in order to learn how to effectively use a lower limb prosthesis. Unfortunately, the process of being fitted a prosthesis can be delayed due to resource constraints and manufacturing times, which delays the rehabilitation process and puts patients at higher risk for functional decline. Preliminary work by our team have shown that our 3D printing system, 3DPrintAbility Devices by NIA (http://niatech.org/), perform at the same level of efficacy as traditionally manufactured prosthetics, which suggests that a digital manufacturing tool-chain is a viable alternative and may be desirable given the time savings involved. In order to lead to improved processes related to prosthesis fitting for adult transtibial amputees, we want to assess the feasibility and acceptability of using 3DPrintAbility sockets in this population. Specifically, we want to determine if: 1) the 3D printing of transtibial prosthetic sockets can provide better quality prosthetic care in regards to cost, timeliness, and accessibility; 2) 3D printed sockets are equivalent in quality to standard thermoplastic preparatory sockets in regards to safety, fit, durability and comfort; and 3) whether a 3D scanning, design and printing process can be integrated into the workflow of current rehab centres. If successful, the findings from this work can provide an innovative approach for facilitating the fitting of a socket for adults with amputation might provide significant savings to the healthcare system by making the process more efficient while optimizing clinical outcomes by allowing patients to begin their rehabilitation sooner

DETAILED DESCRIPTION:
Lower limb amputation (LLA) resulting from trauma or non-traumatic causes is a life altering and often debilitating event that negatively affects many aspects of a person's life, such as their ability to move around the home and community, their physical and mental health. Persons with lower-limb amputation face challenges with activities of daily living and have noted psychosocial issues stemming from poor body image as well as issues of chronic pain from phantom limb syndrome. Further, mortality rates are known to be extremely high, estimated at ~25% at 30 days post amputation and nearly 50% by one year. As the number of LLA continues to rise, this will ultimately lead to an increased demand for services and subsequent greater financial impact to the healthcare system. There are several factors that influence outcomes post-amputation but walking with a prosthesis has been noted to be a central factor influencing quality of life. For instance, greater participation in social experiences is positively associated with mobility outcomes, such as walking distance.

The increasing number of adults requiring care post-amputation is reflected by the large volume of amputee patients receiving care at Sunnybrook Health Sciences Centre's St. John's Rehab (SJR) campus and Sunnybrook's Centre for Independent Living (SCIL). SJR is a tertiary rehabilitation centre with a dedicated in-patient and out-patient amputee care program, and SCIL provides amputee care and prosthetic service at Sunnybrook's Bayview campus. The increased number of LLA creates a high demand for prosthetists as they need to meet with each patient several times to fit them. Due to staffing constraints, there are often delays in prosthetic fitting. With current technologies, it takes one to two weeks from the time Sunnybrook patients are cast and measured until they are fit with their prosthesis. This delay leads to increased rehab length of stay, cost and decreased rehab efficiency.

While a number of companies and individuals are beginning to explore the use of 3Dprinting for mobility prosthetics, few of them have clinical experience beyond a few cases. There are, however, three groups working actively in this space. Vorum Inc., TechMed3D, and Standard Cyborg. All of these are software companies, which are building scanning and design solutions for use in prosthetics. None offers a full single site solution that also includes the printing of definitive devices. Nia Technologies (http://niatech.org/), the technology partner on this project, has developed a full software/hardware tool-chain for prosthetics and has carried out clinical trials at four hospital sites in three developing world countries with pediatric transtibial amputees. For instance, in 2016-2017, Nia worked with clinical partners in Cambodia, Tanzania, and Uganda to study the efficacy and value of 3D PrintAbility to orthopaedic workshops, clinicians, and patients in low-resource countries. The innovation is that the use of Nia technologies enables a 3D model of the residual limb, thereby eliminating the need to use plaster casting and other time consuming processes to manufacture and fit the device. As a result, this technology has the potential to cut time from the assessment to fitting from about 5 days to less than 1.5 days for a prosthetic leg. Preliminary results indicate that the resulting devices were as effective and well-tolerated by patients as traditionally manufactured prostheses. In addition, the use of 3D printing can build on the skills and expertise of physicians and prosthetists since it allows them to minimize time on manual production and maximize time on decisions about device design, fit, and patient care. The innovation being developed in this project leverages Nia's existing work, but focuses it on a specific in-need patient base, namely transtibial amputee rehab adult patients in developed world rehabilitation clinics. This clinical context and patient base is different from the developing world sites where this tool-chain was previously tested. Successful implementation requires adaptation of Nia's tool-chain to support the workflow of clinical staff in adult rehab contexts including physiatrists, physical therapists, and prosthetists.

Patients with a unilateral transtibial amputation (N=20) that are currently in-or out-patients at Sunnybrook - St. John's Rehab (SJR) will be recruited to participate in the evaluation aspect of this quality improvement project. Participants who agree to participate in the quality improvement initiative will be asked by the clinical member within their circle of care to ask if they would be willing to participate in the evaluation aspect collecting data on patient outcomes. Once the participant agrees to be contacted by the research coordinator, they will be given an overview of the study and undergo the informed consent process (Appendix A). The participants will be given one day to provide their consent since the fitting process for a prosthetic starts early in the rehabilitation process. Once consent is received, the participants will receive a 3D printed prosthetic to wear. They will then rate their satisfaction and comfort. Data regarding time and associated cost differences will also be collected.

ELIGIBILITY:
The inclusion criteria for potential patient participants are as follows:

* Current SJR in-patient or out-patient who will be receiving a prosthetic for a LLA;
* Must be medically cleared to participate in the study;
* Fluent in English with no cognitive impairments (ex. clinical depression, brain injury) in order to complete the informed consent process and qualitative interview.

The exclusion criteria for SJR participants includes:

* Those who are not medically cleared to participate in the study
* Have significant cognitive, developmental or language impairments (including a lack of fluency in English)
* Persons who do not have a trans-tibial amputation (i.e., partial foot, transfemoral, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Time to Complete Prosthetic Process - SCIL Form | Immediately post intervention
  Details the clinical, technical, and offsite time for the production and fitting of sockets for amputee patients. The broad categories of tasks captured include: 1) preparation & assessment; 2) shape capture; 3) shape capture to rectification; 4) rectification (modifying); and 5) fabrication. Time will be captured in hours.
Costs Associated with Prosthetic Process - SCIL Form | Immediately post intervention
  The various costs associated with each task (materials, clinician hourly rate, etc.) will also be recorded.

SECONDARY OUTCOMES:
Satisfaction with Socket Ratings | Immediately post intervention
  A numeric scale ranging from 0 (not at all satisfied) to 10 (completely satisfied).
Comfort With Socket Ratings | Immediately post intervention
  A numeric scale to capture socket comfort by patients will also be used (0 = not at all comfortable; 10 = very comfortable).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Mayo, MD; MHSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- St. John's Rehabilitation, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayo AL, Gould S, Cimino SR, Glasford S, Harvey E, Ratto M, Hitzig SL. A qualitative study on stakeholder perceptions of digital prosthetic socket fabrication for transtibial amputations. Prosthet Orthot Int. 2022 Dec 1;46(6):607-613. doi: 10.1097/PXR.0000000000000157. Epub 2022 Jun 7. PMID 36515905